CLINICAL TRIAL: NCT05043155
Title: Strategies to Continue Gynae-oncology Services in the Era of COVID-19 Outbreak: Concerns and Challenges in a Referral Centre in Malaysia
Status: Completed | Type: Observational
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Nirmala Chandralega Kampan, Associate Professor Dr, Universiti Kebangsaan Malaysia Medical Centre
Other Study IDs: UKMMC202105
Record Dates: First submitted 2021-09-13; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Vaccination Refusal; Survivorship
Keywords: Covid19; Vaccination; Gynaeoncology cancer; Cancer survivor
MeSH Terms: conditions — COVID-19; Vaccination Refusal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A short survey involving 100 participants was conducted online to explore the understanding of Covid 19 pandemic impact and importance of vaccination among cancer survivors.

ELIGIBILITY:
Inclusion Criteria: Female cancer survivors or care-taker undergoing national covid 19 vaccine -

Exclusion Criteria: Male, not cancer survivors

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female cancer survivors
Study Population: Female cancer survivors or care-taker undergoing national covid 19 vaccine
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Vaccination refusal | 8 months
  Number of cancer survivors refuse vaccine
Reason for Refusal of Vaccine | 8 months
  Number of cancer survivors refuse vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Dept O&G, UKM Medical Centre, Kuala Lumpur, Malaysia